CLINICAL TRIAL: NCT05230381
Title: Effect of Tranexamic Acid on Intraoperative Blood Loss in Patients Undergoing Brain Meningioma Resections: Study Protocol of a Randomised Controlled Trial
Brief Title: Intravenous Tranexamic Acid Reducing Intraoperative Blood Loss in Huge Meningiomas Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Shu Li, Associate Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022018
Record Dates: First submitted 2022-01-05; First posted 2022-02-08 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Tranexamic Acid; Intraoperative Blood Loss; Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continous infusion group (Active Comparator): Infusion with 20mg/kg tranexamic acid and 5mg/kg/h tranexamic acid.
  Interventions: Drug: Continous infusion
- Single infusion group (Active Comparator): Infusion with 20mg/kg tranexamic acid and same volume 0.9% saline.
  Interventions: Drug: Single infusion
- Placebo group (Placebo Comparator): Infusion with same volume of 0.9% saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Continous infusion — The 20mg/kg tranexamic acid will be diluted into a 50ml syringe and infused followed by 5mg/kg/h tranexamic acid infusion.
  Arms: Continous infusion group
Drug: Single infusion — The 20mg/kg tranexamic acid will be diluted into a 50ml syringe and infused followed by same volume of 0.9% saline.
  Arms: Single infusion group
Drug: Placebo — The 0.9% saline is administered with the same volume at the same speed as the other group.
  Arms: Placebo group

SUMMARY:
Intra-operative blood loss of huge meningioma resection patients on average was over 1000ml. Intra-operative massive hemorrhage was associated with longer hospital of stay, higher expense, and higher mortality. Previous studies indicated intra-operative tranexamic acid infusion would decrease blood loss for cardiac, trauma and obstetric procedures. However, limited researches focusing on the effect of tranexamic acid in neurosurgery population, with heterogenous pathologies. The purpose of this study was to investigate the effect of tranexamic acid on intra-operative blood loss in patients undergoing huge meningioma resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective supratentorial meningioma resection with estimated tumor diameter >5cm on brain image.
* Age between 18-65 years.
* American Society of Anaesthesiologist (ASA) physical status Ⅰ to Ⅲ
* Obtain written informed consent.

Exclusion Criteria:

* Allergic to tranexamic acid.
* History of thrombotic disease.
* History of chronic kidney disease
* Receiving other anticoagulation or antiplatelet treatment.
* Refuse to provide written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Estimated intra-operative blood loss | During surgery
  Estimated intra-operative blood loss is assessed as following formula:collected blood volume in the suction canister (mL) - the volume of flushing (mL) + the volume from gauze tampon (mL).

CONTACTS AND LOCATIONS:
Overall Officials: Shu Li, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu H, Liu M, Zhang X, Ma T, Yang J, Wu Y, Wang J, Li M, Wang J, Zeng M, Zhang L, Jin H, Liu X, Li S, Peng Y. The effect of tranexamic acid on intraoperative blood loss in patients undergoing brain meningioma resections: Study protocol for a randomized controlled trial. PLoS One. 2023 Aug 31;18(8):e0290725. doi: 10.1371/journal.pone.0290725. eCollection 2023. PMID 37651373